CLINICAL TRIAL: NCT03106467
Title: Practical Advantages of Single-port Over Conventional Three-port Laparoscopic Appendectomy in Children: A Randomized Controlled Trial of 400 Cases
Brief Title: Practical Advantages of Single-port Over Three-port Laparoscopic Appendectomy in Children
Acronym: PASTA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hallym University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2014-I124
Record Dates: First submitted 2017-03-27; First posted 2017-04-10 (Actual); Last update posted 2017-04-10 (Actual); Status verified 2017-03

CONDITIONS: Appendicitis
Keywords: appendectomy; laparoscopic; single port; randomized
MeSH Terms: conditions — Appendicitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Single-port laparoscopic appendectomy (Experimental): Single-port laparoscopic appendectomy is performed through single-port which is installed in umbilicus.
  Interventions: Procedure: Single-port laparoscopic appendectomy
- Three-port laparoscopic appendectomy (Active Comparator): Three-port laparoscopic appendectomy is performed using conventional three-port technique which needs two additional ports outside umbilicus in addition to trans-umbilical port
  Interventions: Procedure: Three-port laparoscopic appendectomy

INTERVENTIONS:
Procedure: Single-port laparoscopic appendectomy — Single-port laparoscopic appendectomy: A 1.5 cm skin incision is made inside the umbilicus and single port is introduced through it. The appendix is manipulated by a combination of a 5-mm scope, angulated, and straight instruments. The periappendiceal vessels and appendix are ligated and divided. Specimen is delivered via the transumbilical port. Umbilical fascia and skin are routinely closed.
  Arms: Single-port laparoscopic appendectomy
Procedure: Three-port laparoscopic appendectomy — Three-port laparoscopic appendectomy: CLA requires the introduction of a 30-degree 5-mm or 10-mm rigid scope through a 0.5 - 1.0 cm intra umbilical incision. Two additional 5-mm incisions are made outside umbilicus. Appendectomy is performed in the same manner as described for the SLA above. The umbilical fascia and skin are routinely closed.
  Arms: Three-port laparoscopic appendectomy

SUMMARY:
Despite growing popularity, practical advantages of single-port laparoscopic appendectomy (SLA) over conventional three-port laparoscopic appendectomy (CLA) have yet to be established well in pediatric population.

The investigators designed the randomized controlled trial to clarify practical advantages of SLA over CLA in pediatric population. The investigators compared conversion rate, intra-operative adverse events, operating time, wound complications, intra-abdominal complications, and postoperative hospital stay, changes in postoperative pain severity, and cosmetic outcomes during follow up period between SLA and CLA groups.

DETAILED DESCRIPTION:
Currently the single-port laparoscopic appendectomy (SLA) has gained popularity in pediatric population since it was first reported in 1998 by Esposito et al. Nonetheless, the practical advantages of SLA over conventional three-port laparoscopic appendectomy (CLA) have yet to be established well in pediatric population due to lacking and inconsistent high-level evidences from randomized trials and meta-analysis.

Thus far, in addition to overall postoperative hospital stay, complications such as wound abscess and seroma, intra-abdominal abscess and ileus were reported not to be significantly different between SLA and CLA, while SLA might have taken longer operation time in children and adult. Currently, the advertised benefits on postoperative pain and cosmetic results of SLA incurred suspicion because of heterogeneous data inconsistently supporting SLA from a few RCTs especially in pediatric population. Consequently, a consensus regarding the practical superiority of SLA to CLA has still not been reached particularly in children.

To address this issue, the investigators designed the randomized trial to clarify practical benefits of SLA over CLA in pediatric population. For this, the investigators compared conversion rate, intra-operative adverse events, operating time, wound complications, intra-abdominal complications, and postoperative hospital stay, changes in postoperative pain severity, and cosmetic outcomes during follow up period between SLA and CLA groups. Primary end points were postoperative pain severity and cosmetic satisfaction. Secondary endpoints were intra- and post-operative complication rates, operation time, and postoperative hospital stay.

ELIGIBILITY:
Inclusion Criteria:

* Acute appendicitis was diagnosed in accordance with following clinical, laboratory, and radiographic criteria; history of right lower quadrant pain or periumbilical pain migrating to the right lower quadrant with nausea and/or vomiting. presence direct and indirect tenderness on McBurney's point and/or right lower quadrant guarding. a fever ≥ 38°C and/or white blood cell counts more than 10X10³ cells per mL on complete blood count. diameter of appendix ≥ 6 mm with mural thickening and periappendiceal fat infiltration and/or abdominal fluid collection on appendiceal ultrasonography or abdominopelvic computed tomography.
* Perforated appendicitis: disrupted appendix contour with non-homogenous peritoneal fluid collection in pelvic cavity and/or sub-hepatic space simultaneously with above mentioned clinical, laboratory, and radiographic findings of appendicitis.
* Peri-appendiceal abscess which was preoperatively confirmed by ultrasonographic and/or computed tomographic evidence.

Exclusion Criteria:

* Suspicious diagnosis of appendicitis which was not in accordance with the diagnosis criteria.
* Patients who were subjected to ≥ 2 days of empirical antibiotics therapy for initial symptom prior to diagnosis with acute appendicitis.
* History of coagulation disorders, shock upon admission, previous abdominal surgery, contraindication to general anesthesia, suspected or proven malignancy, and mental illness.

Max Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 400 (Actual)
Dates: Start 2014-11-11 (Actual); Primary Completion 2016-06-30 (Actual); Study Completion 2016-08-31 (Actual)

PRIMARY OUTCOMES:
Post-operative pain (visual analogue scale of pain ranging 0-10) | up to postoperative day 7
  Post-operative pain is measured by visual analogue scale of pain ranging 0-10.
Cosmetic satisfaction (visual analogue scale of cosmetic result ranging 1-10) | at postoperative 12 months
  Cosmetic satisfaction is measured by visual analogue scale of cosmetic result ranging 1-10.

SECONDARY OUTCOMES:
Wound complications | up to postoperative 3 months
  Wound complications include port site seroma collection and abscess formation.
Intra-abdominal complications | up to postoperative 3 months
  Intra-abdominal complications include radiologically confirmed bowel ileus or peritoneal abscess formation.
Operation time | on postoperative day 1
  OT is defined as the duration of surgery, from skin incision to application of wound dressing.
Post-operative hospital stay | at postoperative 2 weeks
  Post-operative hospital stay is the days between a day after surgery and discharge. Operation day is considered as day 0.

CONTACTS AND LOCATIONS:
Overall Officials: Soo Min Ahn, MD, Principal Investigator — Division of Pediatric Surgery, Hallym University Sacred Heart Hospital
Locations (1):
- Hallym University Sacred Heart Hospital, Anyang-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: Yes